CLINICAL TRIAL: NCT03676582
Title: The AspiRATE Study: a Proof-of-concept Assessment of a Novel Intervention to Acoustically Detect Silent Aspiration in Patients With Acquired Dysphagia.
Brief Title: AspiRATE: Novel Intervention to Acoustically Detect Silent Aspiration in Acquired Dysphagia.
Acronym: AspiRATE
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Sponsor
Other Study IDs: STH19484
Record Dates: First submitted 2018-09-14; First posted 2018-09-18 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Dysphagia, Oropharyngeal
Keywords: swallowing disorders; instrumental swallow assessment; acoustic analysis; respiratory changes
MeSH Terms: conditions — Deglutition Disorders | interventions — Oximetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Acoustic analysis plus pulse oximetry — Acoustic analysis plus pulse oximetry

SUMMARY:
This study will investigate whether silent aspiration during swallowing can reliably be detected using acoustic signal processing plus pulse oximetry.

DETAILED DESCRIPTION:
This proof of concept trial, involving original research from a multicentre, multidisciplinary team, aims to establish whether silent aspiration can be detected in patients with dysphagia (swallowing difficulties), using a microphone array attached to the neck (to capture acoustic respiratory changes), pulse oximetry (to detect reduction in blood oxygen levels) and respiratory rate analysis, with data combined and analysed via post-capture signal processing techniques.

The project aims to develop equipment and signal processing algorithms to a point where a novel intervention has been established that allows semi-automated detection of safe versus unsafe (aspiration) swallows. The intervention will be trialled in patients with dysphagia within standard videofluoroscopy clinics under clinical supervision. There will be on-going development of the intervention and signal processing algorithms during this process. Public and patient involvement work will feed back into the design process.

If the intervention performs successfully in this proof-of-concept study, the investigators aim to proceed to a larger clinical trial to determine its sensitivity and specificity as a screening tool for aspiration, before final development into a commercial product.

ELIGIBILITY:
Inclusion Criteria:

* Dysphagia ± aspiration,
* age 18 and above

Exclusion Criteria:

* Not competent for consent,
* previous neck surgery (not including thyroid surgery)
* cervical skin infection or defect
* pregnant (or unknown pregnancy status).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults over the age of 18 years with acquired dysphagia
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Pownall, Ph.D, Principal Investigator — Sheffield Teaching Hospitals NHS FT
Locations (1):
- Sheffield Teaching Hospitals NHS FT, Sheffield, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
As this is a proof of concept study, ethical approval has been secured for sharing of anonymised patient data with research study named collaborators for input advice on advanced data analysis. This is included on patient information and recruitment processes.

RESULTS

PARTICIPANT FLOW:
Groups:
- Stroke Patients: Stroke patients - with acquired dysphagia
Period: Overall Study
Arm/Group | Stroke Patients
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with acquired dysphagia
Arm/Group | Stroke Patients
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 25

OUTCOME MEASURES:

1. Primary Outcome: Presence or Absence of Aspiration
Description: Presence or absence of matter passing between or below the vocal cords during swallowing, particularly in the absence of cough reflex stimulation - novel intervention to acoustically detect silent aspiration in patients
Time Frame: 1 hour
Population: Stroke patients with acquired dysphagia undergoing videofluoroscopy
Measure: Number; unit: swallowing events with aspiration
Groups:
- Swallowing Events: Swallowing events of Stroke patients - with acquired dysphagia
Arm/Group | Swallowing Events
Number analyzed (Participants) | 16
swallowing events with aspiration | 42

ADVERSE EVENTS:
Time Frame: From informed consent to study completion (Time frame per participant: up to 1 day)
Description: As per protocol
Arm/Group | Stroke Patients
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

LIMITATIONS AND CAVEATS:
Some swallowing events had to be excluded because of background noise in the recording.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT03676582/Prot_000.pdf